CLINICAL TRIAL: NCT04173780
Title: Topical 0.01% Atropine for the Control of Fast Progressing Myopia
Acronym: Myopie-STOP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7343
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Myopia Progressing; Childhood
Keywords: Myopia (Progressing); Childhood; Atropine 0,01%
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atropine 0.01% (Experimental)
  Interventions: Drug: Atropine 0.01%
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atropine 0.01% — 1 drop per day in both eyes for 1 year
  Arms: Atropine 0.01%
Drug: Placebo — 1 drop per day in both eyes for 1 year
  Arms: Placebo

SUMMARY:
Myopia prevalence has dramatically increased worldwide in recent years in the general population and among children. Progressive myopia increases gradually with growth until the age of 20-25 years. At the same time, there is a remarkable increase in the prevalence of severe myopia (more than -6 diopters). Severe myopia is associated with many complications, which can lead to blindness. There is thus an increase in the number of myopic patients in general, and severe myopic patients in particular.

The management of myopia and its complications is therefore a major public health issue.

All the means likely to slow the evolution of myopia (thus to limit the prevalence of strong myopia) must be developed to limit the consequences. 0.01% Atropine seems to be a drug with a great interest to slow down the progression of myopia.

The aim of the present study is to evaluate the efficacy at 1 year of 0.01% atropine (1 drop per day administered for 1 year) on the reduction of fast progressing myopia in children aged 4 to 12, compared to a control group (instillation of a placebo).

ELIGIBILITY:
Inclusion Criteria:

Children from 4 to 12 years

* Myopia from -1 to -6
* Fast progressing myopia (>0.75 diopter / year)
* Informed consent obtained

Exclusion Criteria:

Astigmatism > 1.5 diopters

* Anisometropia > 2 diopters
* Concomitant pathology of anterior or posterior segments
* Other ocular diseases (Ocular inflammation, strabismus …)
* Atropine hypersensitivity or allergy

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Myopia in spherical diopters | 12 months
  Automatic measurement of myopia in spherical diopters under cycloplegia
Myopia in spherical diopters | 9 months
  Automatic measurement of myopia in spherical diopters under cycloplegia
Myopia in spherical diopters | 6 months
  Automatic measurement of myopia in spherical diopters under cycloplegia
Myopia in spherical diopters | 3 months
  Automatic measurement of myopia in spherical diopters under cycloplegia

SECONDARY OUTCOMES:
Axial length | 12 months
Axial length | 6 months
Axial length | 3 months
Axial length | 9 months
Adverse events | 12 months
Adverse events | 9 months
Adverse events | 6 months
Adverse events | 3 months
Quality of life questionnaire | 12 months
Quality of life questionnaire | 9 months
Quality of life questionnaire | 6 months
Quality of life questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud SAUER, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- CHU de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No